CLINICAL TRIAL: NCT06956612
Title: Evaluating the Impact of Various Dietary Nitrate Supplementation Forms on Microbiological Markers of Oral Health and Acceptability Among Adult Participants
Brief Title: Evaluating the Impact of Various Dietary Nitrate Supplements on Oral Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shatha Alhulaefi (Other)
Collaborators: Northumbria University (Other); Edith Cowan University (Other); University of the West of Scotland (Other)
Responsible Party: Sponsor-Investigator, Shatha Alhulaefi, Doctoral Researcher, Newcastle University
Organization: Newcastle University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2966/53998
Record Dates: First submitted 2025-04-24; First posted 2025-05-04 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Oral Health; Dietary Nitrate
Keywords: Dietary nitrate; oral health; salivary acidity; oral microbiome

STUDY DESIGN:
Who Masked: Participant
Masking Description: This study will use a single-blind design, where the participants will not know whether they receive the real supplement or the placebo. Participants will be told they might receive either crystals or juice, but they won't know whether it's an active supplement or a placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Daily supplementation with 70 ml nitrate-depleted Beet It Sport Shots, James White Ltd (~0mg dietary nitrate)
  Interventions: Dietary Supplement: Control (Placebo comparator)
- Juice (Active Comparator): Daily supplementation with 70 ml Beet It Sport Shots, James White Ltd (~400mg nitrate).
  Interventions: Dietary Supplement: Juice (Active comparator)
- Crystals (Experimental): Daily supplementation with 20g Beet It Sport Crystals, James White Ltd (~400mg nitrate).
  Interventions: Dietary Supplement: Crystals (Experimental)

INTERVENTIONS:
Dietary Supplement: Control (Placebo comparator) — The control group will consume a placebo supplement, entirely free of nitrate, in the form of juice (70 ml) for four weeks while maintaining their habitual diet.
  Arms: Control
Dietary Supplement: Juice (Active comparator) — The juice group will consume a beetroot supplement enriched with ~400 mg of nitrate in juice form (70 ml) for four weeks while maintaining their habitual diet.
  Arms: Juice
Dietary Supplement: Crystals (Experimental) — The crystals group will consume a beetroot supplement enriched with ~400 mg of nitrate in crystals form (20g) for four weeks while maintaining their habitual diet.
  Arms: Crystals

SUMMARY:
This study aims to investigate the effects of different dietary nitrate supplements, versus placebo, on microbiological and immunological markers associated with oral health in people aged 18-65 years.

The main research questions are:

* How do different dietary nitrate supplements (beetroot crystals vs. beetroot juice) affect oral health markers, including salivary pH and oral microbiome composition?
* What is the acceptability and ease of integrating one of dietary nitrate supplements, made from beetroot but processed as freeze dried crystals or juice, into the daily diet?

To answer these questions, the study will compare results from three groups of participants, who will be randomly assigned to one of the following study arms:

Group 1: The control group will consume a placebo beetroot supplement completely free of nitrate in juice form.

Group 2: The beetroot juice group will consume a beetroot supplement standardised to contain ~ 400 mg of nitrate in juice form.

Group 3: The beetroot crystals group will consume a beetroot supplement standardised to contain ~400 mg of nitrate in freeze dried crystal form.

The study will follow a randomised, single-blind, placebo-controlled, parallel design, and the intervention will last for four weeks. Data will be collected by providing pre- and post-intervention saliva samples tongue swabs, and various questionnaires will be completed at baseline and at the end of the study. In addition, at the end of the second week of the intervention period, participants will be asked to collect a saliva sample over three consecutive days at home.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged 18 - 65 years.

Exclusion Criteria:

* Aged less than 18 or more than 65 years old.
* Current smoking
* Alcohol consumption of greater than14 units per week.
* Diagnosis of a chronic disease (e.g., cardiovascular disease, diabetes, cancer, or gastrointestinal disorders), including oral diseases.
* Use of antibiotics within the past three months or medications/nutritional supplements that may affect the oral cavity (e.g., prebiotics, probiotics, or hormone replacement therapy).
* Regular use of antibacterial mouthwash or xylitol-containing products (e.g., gum or toothpaste) or the use of proton pump inhibitors.
* Presence of braces/invisalign or dentures.
* Known allergy to any food, including beets
* Adherence to dietary restrictions (e.g., weight loss diet)
* Eating disorders that may limit participation in the study.
* Currently pregnant, breastfeeding or trying to become pregnant.
* Participation in other studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Saliva pH | 4 weeks
  Prior to and following the intervention, participants will provide an unstimulated saliva sample for pH measurement. The pH of each saliva sample will be measured using a pre-calibrated pH meter (±0.01 pH accuracy). Measurements will be performed in three independent replicates for each sample, with the three values recorded and then averaged. This average is used for the final pH value of the sample, helping to reduce the influence of random errors and improve the accuracy and reliability of the results. The device is recalibrated prior to measurements using standard calibration solutions to ensure accurate readings.
Oral microbiome | 4 weeks
  Prior to and following the intervention, participants will provide unstimulated saliva and tongue swab samples. DNA will be extracted from both the saliva and tongue swab samples, and 16S rRNA sequencing will be performed to identify and quantify changes in the oral microbiome.

SECONDARY OUTCOMES:
Salivary nitrate/ nitrite concentrations | 4 weeks
  Prior to and following the intervention, participants will provide an unstimulated saliva sample to determine saliva nitrate and nitrite levels using ozone-based chemiluminescence. Home-collected saliva samples will also be analysed for three consecutive days to ensure compliance.
Saliva flow rate | 4 weeks
  Participants will provide an unstimulated saliva sample prior to and following the intervention. The saliva volume collected (in mL) will be divided by the time taken (in min) to obtain the flow rate in ml/min.
Salivary biomarkers | 4 weeks
  Participants will provide an unstimulated saliva sample prior to and following the intervention. If sufficient sample volume is available, exploratory analysis of salivary biomarkers related to inflammation may be considered.
Dry mouth severity (Xerostomia) | 4 weeks
  The impact of the study interventions on dry mouth symptom severity pre- and post-intervention will be assessed using the Summated Xerostomia Inventory-Dutch Version (SXI-D) questionnaire (Thomson et al., 2011), which has been validated in clinical and epidemiological research. Participants will provide information about their oral symptoms over the previous four weeks (e.g., feeling dry mouth or difficulty eating dry foods). Participants will be asked to select one of three options, each of which is associated with a score (Never (1); Occasionally (2) and Often, (3)). The SXI-D score range is 5-15, with higher scores indicating more severe dry mouth.
Oral hygiene behaviours | 4 weeks
  Participants will provide information on their oral hygiene behaviours before and after the intervention using the Oral Hygiene Behaviour Index questionnaire (Buunk-Werkhoven et al., 2011). The score ranges from 0 to 16, with a high total score indicating a high level of oral hygiene practices.
Dietary nitrate intake assessment | 4 weeks
  Before and after the intervention, participants will provide information about their intake of nitrate containing foods through a validated digital food frequency questionnaire(McMahon et al., 2023).
Intervention acceptability | 4 weeks
  The acceptability of the interventions will be assessed after the study is completed through a questionnaire designed to measure acceptability dimensions according to the Theoretical Framework of Acceptability (Sekhon et al., 2017), using a 5-point Likert scale to assess different aspects such as overall acceptability, palatability, and ease of use.
Participant Compliance | 4 weeks
  Compliance will be assessed using a participant-completed compliance log over a 4-week period. Participants will be asked to record:
  * The date and time of supplement intake.
  * How it was consumed. Additionally, any unused supplement sachets/bottles will be collected at the final visit to help estimate adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Shannon, PhD, Principal Investigator — Newcastle University; Anthony Watson, PhD, Principal Investigator — Newcastle University; Sheena Ramsay, PhD, Principal Investigator — Newcastle University
Locations (1):
- Newcastle University, Newcastle upon Tyne, Tyne and Wear NE2 4HH, Newcastle, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided